CLINICAL TRIAL: NCT05189938
Title: HbA1c Variation Study
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-RES-21212
Record Dates: First submitted 2021-12-20; First posted 2022-01-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus
Keywords: Professional FreeStyle Libre Flash Glucose Monitoring System; HBA1C
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HBA1c data and glucose levels — All subjects will wear the professional FreeStyle Libre Pro for glucose data and HbA1c data will be collected at different time points over the participation period.

SUMMARY:
To evaluate the relationship between glycated hemoglobin (HbA1c) and average glucose levels using continuous glucose monitoring.

DETAILED DESCRIPTION:
This is a non-pivotal , non-randomized, single-arm, multi-center, prospective, non-significant risk study to evaluate the relationship between glycated hemoglobin (HbA1c) and average glucose levels. Up to approximately 600 subjects will be enrolled who will have fourteen (14) study visits over the course of approximately six (6) months. During each visit the subject will have blood samples drawn for documentation of their HbA1c level. Subjects will also be required to wear Professional FreeStyle Libre Flash Glucose Monitoring System(s) to record blood glucose levels through the duration of the study. During Visits 1 and 14, Venous sample for CBC, biochemistry, haemoglobinopathy screen, hematology, liver function and iron panels will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have type 1 or type 2 diabetes.
2. Subject is at least 4 years old.
3. Point-of-care (POC) HbA1C of 3.0%-15.5% (9 mmol/mol - 146 mmol/mol)
4. Subject must be able to read and understand English.
5. In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
6. Subject must be available to participate in all study visits.
7. Subject must be willing and able to provide written signed and dated informed consent.
8. Subjects age 4 - 17: Parent or guardian must be willing and able to provide written signed and dated informed consent.
9. Subjects age 11 - 17 Subject must be willing and able to provide written signed and dated informed assent.

   Exclusion Criteria:
10. Subject is currently undergoing dialysis or planning to receive dialysis during the course of the study
11. History of blood transfusion in the last 3 months or planned blood transfusion during the course of the study.
12. Subject is currently planning to undergo a major medical intervention expected to significantly alter red cell life span, i.e. chemotherapy, major surgery requiring blood transfusions, etc.
13. Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
14. Subjects age 18 and older: Subject is known to be pregnant, attempting to conceive or is not willing and able to practice birth control during the study duration study (applicable to female subjects only). Subjects age 17 and younger: Subject is known to be pregnant at the time of study enrollment or is planning to become pregnant during the study (applicable to female subjects only).
15. Subject has extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements. Such conditions include, but are not limited to extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, dermatitis herpetiformis, skin lesions, redness, infection or edema.
16. Subject has a pacemaker or any other neurostimulators.
17. Subject has concomitant medical condition which, in the opinion of the investigator, could present a risk to the safety or welfare of the subject or study staff.
18. Subject is currently participating in another interventional clinical trial.
19. Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with type 1 or 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 488 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Establish a relationship between laboratory-derived HbA1c and average glucose levels | six (6) months
  This is an observational data collection study, where the goal is to gather data to establish the relationship between laboratory-derived HbA1c and average glucose levels.

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara A Karinka, PhD, Study Director — Abbott Diabetes Care
Locations (22):
- United States (8):
  - Excellence Research and Medical, Miami Gardens, Florida
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Billings Clinic, Billings, Montana
  - Albuquerque Neuroscience Inc., Albuquerque, New Mexico
  - Anmed Health Internal Medicine Associates, Anderson, South Carolina
  - Prime Revival Research Institute, Flower Mound, Texas
  - Eastside Research Associates, Redmond, Washington
  - Rainier Clinical Research Center, Renton, Washington
- United Kingdom (14):
  - University Hospital Birmingham, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Royal Derby Hospital, Derby
  - Edinburgh Royal Infirmary, Edinburgh
  - Northwick Park Hospital, Harrow
  - Hull Royal Infirmary, Hull
  - St James University Hospital, Leeds
  - Leicester General Hospital, Leicester
  - Manchester Royal Infirmary, Manchester
  - Nottingham Children's Hospital & Queen's Medical Centre, Nottingham
  - Royal Berkshire Hospital, Reading
  - Northern General Hospital, Sheffield
  - Ealing Hospital, Southall
  - The Royal London Hospital, Whitechapel